CLINICAL TRIAL: NCT05328999
Title: Fertility and the Microbiome: an Observational Study and Randomized Placebo Controlled Double-blind Pilot Trial
Brief Title: Fertility and the Microbiome
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: Fertilitom
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Subfertility; Asthenozoospermia
MeSH Terms: conditions — Infertility; Asthenozoospermia | interventions — Probiotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oral swabs, vaginal swabs, uterine swabs, cervical swabs, urine, ejaculate, stool samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subfertile patients: Males and females between 18 and 50 years of age with subfertility presenting at the fertility center at the Medical University of Graz.
- Subfertile males with elevated DNA fragmentation index and asthenozoospermia: Males between 18 and 50 years of age with elevated DNA fragmentation index and asthenozoospermia presenting at the fertility center at the Medical University of Graz.
  Interventions: Dietary Supplement: Probiotics (Omnibiotic (R))

INTERVENTIONS:
Dietary Supplement: Probiotics (Omnibiotic (R)) — As intervention in the randomized placebo controlled double blind trial, 30 males will receive either probiotics or placebo once daily for 3 months. Sperm count and microbiome analysis before and after intervention will be performed.
  Groups: Subfertile males with elevated DNA fragmentation index and asthenozoospermia

SUMMARY:
With this study, the investigators want to investigate the microbiome and human papilloma virus (HPV) status of couples with subfertility. The investigators want to gain information about association of female and male microbiome and its impact on fertility. HPV prevalence is high, and its impact on fertility has not been studied intensively. The investigators want to find out whether there is an association between HPV status and subfertility, vaginal and seminal microbiome and HPV status and the prevalence among our subfertile couples.

As part of this study, the investigators will perform a randomized placebo controlled double blind pilot study to investigate the association between altered sperm quality (impaired motility and elevated DNA fragmentation index), the seminal microbiome and whether intake of probiotics alters these parameters.

DETAILED DESCRIPTION:
Observational study:

The investigators will include 150 couples within 24 months and will take samples of oral, urinary, stool, vaginal, uterine and seminal microbiome and cervical as well as seminal samples for HPV analysis. Further, the investigators will test for other sexually transmittable diseases, hormone status and metabolic status. Time to pregnancy, pregnancy rate and live birth rate will be evaluated.

Placebo controlled double blind randomized controlled trial:

30 subfertile men (Asthenozoospermia, elevated DNA fragmentation index) will be randomized in to two groups: Placebo or Probiotics for 3 months daily. Before and after these 3 months, sperm count microbiome analysis and HPV analysis will be performed to find possible associations with intake of probiotics.

ELIGIBILITY:
Inclusion Criteria:

* Couples (Males and females) with subfertility, primary or secondary infertility, or recurrent pregnancy loss.

Exclusion Criteria:

* unable to consent
* diseases or conditions that might impact investigation
* intake of probiotics, antibiotics within last 3 months
* intake of nutritional supplements
* chemo therapy or radiation therapy
* excess alcohol intake
* smoking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Couples (Males and females) with subfertility, primary or secundary infertility, or recurrent pregnancy loss.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2025-04-11 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Seminal microbiome | 3 months
  16S-RNA sequencing; shotgun metagenomic sequencing
Vaginal microbiome | 1 month
  16S-RNA sequencing; shotgun metagenomic sequencing
Uterine microbiome | 1 month
  16S-RNA sequencing; shotgun metagenomic sequencing
DNA-Fragmentation index | 3 months
  Rate of sperm with elevated DNA Fragmentation index

SECONDARY OUTCOMES:
Hormone status of males and females - LH (Luteinizing hormone) | 3 months
  LH status
Hormone status of males and females - FSH (follicle stimulating hormone) | 3 months
  FSH status
Hormone status of males and females - Testosterone status | 3 months
  Testosterone status
Hormone status of males and females - free Testosterone | 3 months
  free Testosterone status
Hormone status of males and females - Androstenedione | 3 months
  Androstenedione status
Hormone status of males and females - AMH (Anti-Müllerian hormone) | 3 months
  AMH status
Hormone status of males and females - DHEAS (dehydroepiandrosterone sulphate) | 3 months
  DHEAS status
Hormone status of males and females - 25(OH)Vitamin D | 3 months
  25(OH)Vitamin D status
Hormone status of males and females - TSH (thyroid-stimulating hormone) | 3 months
  TSH status
Hormone status of males and females - fT3 (free Triiodothyronine) | 3 months
  fT3 Status
Hormone status of males and females - freeThyroxine (fT4) | 3 months
  fT4 status
HPV Status | 3 months
  HPV PCR analysis
stool microbiome | 3 months
  16S-RNA sequencing; shotgun metagenomic sequencing
oral microbiome | 3 months
  16S-RNA sequencing; shotgun metagenomic sequencing
Cortisol in Saliva | 3 months
  cortisol analysis in saliva of females and males
Amylase in Saliva | 3 months
  amylase analysis in saliva of females and males
Metabolic parameters - Omega 3 | 3 months
  Omega 3
Metabolic parameters - Omega 6 | 3 months
  Omega 6
Metabolic parameters - low density lipoprotein | 3 months
  low density lipoprotein
Metabolic parameters - high density lipoprotein | 3 months
  high density lipoprotein
Metabolic parameters - triglycerides | 3 months
  triglycerides
Metabolic parameters - LipoproteinA | 3 months
  LipoproteinA
Time to pregnancy | 24 months
  Time until clinical pregnancy is achieved
pregnancy rate | 24 months
  rate of clinical pregnancies
live birth rate | 24 months
  follow up of pregnancies and their outcome
Presence of sexual transmittable diseases | 3 months
  HBV, HCV, HIV, Syphilis, Chlamydia, Gardnerella, Trichomonas
Sperm count | 3 months
  Motility, concentration, morphology

CONTACTS AND LOCATIONS:
Overall Officials: Martina Kollmann, PD Dr., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jersoviene V, Gudleviciene Z, Rimiene J, Butkauskas D. Human Papillomavirus and Infertility. Medicina (Kaunas). 2019 Jul 15;55(7):377. doi: 10.3390/medicina55070377. PMID 31311196
- [Background] Brusselaers N, Shrestha S, van de Wijgert J, Verstraelen H. Vaginal dysbiosis and the risk of human papillomavirus and cervical cancer: systematic review and meta-analysis. Am J Obstet Gynecol. 2019 Jul;221(1):9-18.e8. doi: 10.1016/j.ajog.2018.12.011. Epub 2018 Dec 12. PMID 30550767
- [Background] Koedooder R, Singer M, Schoenmakers S, Savelkoul PHM, Morre SA, de Jonge JD, Poort L, Cuypers WJSS, Beckers NGM, Broekmans FJM, Cohlen BJ, den Hartog JE, Fleischer K, Lambalk CB, Smeenk JMJS, Budding AE, Laven JSE. The vaginal microbiome as a predictor for outcome of in vitro fertilization with or without intracytoplasmic sperm injection: a prospective study. Hum Reprod. 2019 Jun 4;34(6):1042-1054. doi: 10.1093/humrep/dez065. PMID 31119299
- [Background] Depuydt CE, Donders GGG, Verstraete L, Vanden Broeck D, Beert JFA, Salembier G, Bosmans E, Ombelet W. Infectious human papillomavirus virions in semen reduce clinical pregnancy rates in women undergoing intrauterine insemination. Fertil Steril. 2019 Jun;111(6):1135-1144. doi: 10.1016/j.fertnstert.2019.02.002. Epub 2019 Apr 17. PMID 31005311
- [Background] Baud D, Pattaroni C, Vulliemoz N, Castella V, Marsland BJ, Stojanov M. Sperm Microbiota and Its Impact on Semen Parameters. Front Microbiol. 2019 Feb 12;10:234. doi: 10.3389/fmicb.2019.00234. eCollection 2019. PMID 30809218
- [Background] Koedooder R, Singer M, Schoenmakers S, Savelkoul PHM, Morre SA, de Jonge JD, Poort L, Cuypers WSS, Budding AE, Laven JSE; ReceptIVFity study group. The ReceptIVFity cohort study protocol to validate the urogenital microbiome as predictor for IVF or IVF/ICSI outcome. Reprod Health. 2018 Dec 7;15(1):202. doi: 10.1186/s12978-018-0653-x. PMID 30526664
- [Background] Depuydt CE, Donders G, Verstraete L, Vanden Broeck D, Beert J, Salembier G, Bosmans E, DhontT N, Van Der Auwera I, Vandenborne K, Ombelet W. Time has come to include Human Papillomavirus (HPV) testing in sperm donor banks. Facts Views Vis Obgyn. 2018 Dec;10(4):201-205. PMID 31367292
- [Background] Xiong YQ, Chen YX, Cheng MJ, He WQ, Chen Q. The risk of human papillomavirus infection for male fertility abnormality: a meta-analysis. Asian J Androl. 2018 Sep-Oct;20(5):493-497. doi: 10.4103/aja.aja_77_17. PMID 29623908
- [Background] Moreno I, Simon C. Relevance of assessing the uterine microbiota in infertility. Fertil Steril. 2018 Aug;110(3):337-343. doi: 10.1016/j.fertnstert.2018.04.041. PMID 30098680
- [Background] Simon C. Introduction: Do microbes in the female reproductive function matter? Fertil Steril. 2018 Aug;110(3):325-326. doi: 10.1016/j.fertnstert.2018.06.041. Epub 2018 Jul 20. PMID 30037698